CLINICAL TRIAL: NCT04375358
Title: Creatinine Clearance as a Predictor of Successful Withdrawl of Continuous Renal Replacement Therapy in Intensive Care
Acronym: STOP EERc
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: NGUYEN 2018
Record Dates: First submitted 2020-04-27; First posted 2020-05-05 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Dialysis Withdrawal; Creatinine Clearance
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood and urine samples — To measure the clearance of creatinine, urea, potassium, magnesium, sodium, chlorine...

SUMMARY:
Acute renal failure is a common complication in patients admitted to intensive care. Due to the increasing incidence of acute renal failure, the use of Continuous Renal Replacement Therapy (CRRT) is on the rise in the intensive care unit. The use of CRRT exposes patients to some complications (bleeding, hemodynamic instability, antibiotic underdosing, malnutrition and infections), justifying the importance of optimizing the quality and reliability of this technique. Renal function is classically assessed by diuresis and creatinine. Creatinine clearance is an indirect measure of glomerular filtration rate. Measuring creatinine clearance is a simple, accessible and relatively inexpensive method. Traditionally, clreatinine clearance has required 24-hour urine collection. However, it has been shown that two-hour urine collection is also an accurate tool.

There is little information and few recommendations as to when to discontinue CRRT. A predictive index for the withdrawal of CRRT would reduce the duration of treatment, reduce complications and costs, and speed up patient rehabilitation.

Various parameters have been described as tools for deciding when to stop dialysis: diuresis before stopping CRRT, urine and blood creatinine, daily urinary urea excretion, and sodium and water balance. Among these factors, urine output and creatinine appear to be promising predictive factors. The measurement of creatinine clearance combines these two factors and can therefore be a good tool for predicting the return of adequate renal function. Retrospective work carried out by Fröhlich et al in 2012 suggested that creatinine clearance measured over 2 hours could be a good marker for successful withdrawal.

The hypothesis of the study is that creatinine clearance measured over 2 hours after stopping CRRT is be predictive of the success of the withdrawal from this type of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis for AKI with minimum 12 hours of continuous renal replacement therapy (CVVH-CVVHD)
* Patient in whom dialysis withdrawal is being considered
* Patients over 18 years of age

Exclusion Criteria:

* Pre-existing chronic end-stage renal failure on chronic dialysis
* Extrarenal purification during hospitalization prior to admission to intensive care unit
* Inability to assess the primary outcome
* Kidney Transplantation
* Pregnant Women
* Person not affiliated to a national health insurance
* Decision to limit or stop therapy
* Isolated hyperkalemia
* Refusal of patient participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
creatinine clearance over 2 hours | Through study completion, an average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France